CLINICAL TRIAL: NCT07019467
Title: The Effect of Bed Bath Given to Intensive Care Unit Patients With Auditory Hypnosis on Physiological and Comfort Parameters: a Randomized Controlled Experimental Study
Brief Title: Bed Bath With Auditory Hypnosis on ICU Patients
Acronym: RCS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Banu Terzi (Other)
Responsible Party: Sponsor-Investigator, Banu Terzi, Associate Professor, Akdeniz University
Organization: Akdeniz University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Bntz2025; Bath2025 (Other: Akdeniz University)
Record Dates: First submitted 2025-05-19; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Critical Care
Keywords: auditory hypnosis; bed bath; comfort; critical ill patients; ICU; physiological parameters

STUDY DESIGN:
Intervention Model Description: Experimental, randomised controlled, single-blind study
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomised
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bed bath with auditory hypnosis (Experimental): In the bed bath protocol accompanied by auditory hypnosis; An audio recording with 30-60 minutes of auditory hypnosis content specific to the ICU patient will be prepared with the support of an expert hypnotherapist. This audio recording will include the following messages: - The purpose of the bed bath, - Procedures to be performed during the bed bath, - Benefits of the bed bath, - Feeling safe during the bed bath, - Improvement of physiological parameters and comfort level after the bed bath.
  Interventions: Other: Bed Bath With Auditory Hypnosis
- Control Group (No Intervention): In this study, the control group will receive standard bed bath.

INTERVENTIONS:
Other: Bed Bath With Auditory Hypnosis — In the bed bath protocol accompanied by audio suggestion, a 30-60 minute audio recording containing audio suggestions specific to the ICU patient will be prepared with the support of a specialist hypnotherapist. This audio recording will include the following messages: - The purpose of the bed bath, - Procedures to be performed during the bed bath, - The benefits of the bed bath, - Feeling safe during the bed bath, - Improvement in physiological parameters and comfort levels after the bed bath.
  While it is noted that auditory suggestion typically lasts 30-60 minutes, even a 15-minute auditory suggestion has been reported to provide benefits.
  Arms: Bed bath with auditory hypnosis

SUMMARY:
Intensive care units (ICUs) are specialized units where complex life-saving treatment and care activities are performed. Due to the treatment procedures performed in these specialized units, a large number of tools/equipment/devices/cables (endotracheal tubes, monitor cables, hemodialysis machines, mechanical ventilation, etc.) are placed on critically ill patients. These treatment devices restrict the movement of patients, creating obstacles to the independent performance of basic human needs such as personal hygiene. One of the individual hygiene practices frequently applied in ICUs is bed bathing. The application of bed bathing in ICUs varies according to institutional and clinical policies. In addition to its beneficial effects such as preventing infection, accelerating blood circulation, providing comfort and relaxation, etc., bed bathing also carries the risk of having a negative effect on physiological parameters. Eliminating or minimizing this risk is one of the primary care objectives of intensive care nurses. In this regard, it is crucial that bed baths, which are considered a routine nursing activity in ICUs, are performed in accordance with specific standards and protocols. In recent years, there has been an increase in the use of certain non-pharmacological care interventions in ICUs. One such intervention is auditory suggestion. Auditory suggestion refers to messages delivered through hearing to facilitate the adoption of specific thoughts, feelings, or behaviors. This method includes music, verbal suggestion, nature sounds, and other auditory stimuli that are believed to have the potential to influence the subconscious. In recent years, auditory suggestion has been integrated into the treatment processes of critically ill patients, particularly in intensive care units. This method is applied to reduce patients' stress, control pain, and support hemodynamic stability. Research has provided strong evidence supporting the physiological and psychological effects of auditory suggestion on both adult and pediatric patients. On the other hand, maintaining the patient's physiological parameters under control and increasing their comfort level while administering bed baths in the ICU are desired outcomes of nursing care. Based on this, the study was designed as a randomized controlled trial to investigate the effects of bed baths administered with auditory suggestion on physiological and comfort parameters in intensive care patients. The study, which will be conducted with a total of 66 ICU patients meeting the sample selection criteria, will apply the "bed bath protocol with auditory suggestion" to the study group and routine bed baths to the control group (only once). The study data will be collected using the "Patient Information Form" and the "Physiological and Comfort Parameters Monitoring Form" (data from the form will be collected and recorded before the bath, immediately after the bath, and 30 minutes after the bath). The study data will be analyzed using appropriate statistical methods.

DETAILED DESCRIPTION:
Intensive care units (ICU) are specialized units where complex life-saving treatment and care activities are performed. Due to the treatment interventions applied in these special units, a large number of tools/equipment/devices/cables (intubation tube, monitor cables, hemodialysis device, mechanical ventilation, etc.) are placed in critically ill patients. These treatment equipments restrict the movement of patients and hinder the independent fulfillment of the most basic human needs such as personal hygiene. One of the most common individual hygiene practices in ICUs is bed bathing. At the same time, in addition to the beneficial effects of bed bathing such as preventing infection, accelerating blood circulation, providing comfort and relaxation, etc., there is also a risk of negative effects on physiological parameters. Elimination or minimization of this risk is one of the primary care-giving goals of the intensive care nurse.

Considering the duties, authorities and responsibilities of intensive care nurses, ensuring the safety and comfort of the critical patient in the ICU should be the primary goal of the nurse. In this direction, some non-pharmacological applications can be utilized to prevent the risk of deterioration in the patient's physiological parameters and to increase his/her comfort during bed bathing, which is frequently applied to critically ill patients in the ICU and seen as an ordinary procedure.

One of these applications, the effects of which have been investigated on critically ill patients in ICU in recent years, is auditory suggestion. Auditory suggestion refers to verbal or auditory messages given through hearing to facilitate individuals to adopt certain thoughts, feelings or behaviors. This method includes music, verbal suggestion, nature sounds and other auditory stimuli that are thought to have the potential to influence the subconscious mind.

Recent studies have shown that auditory suggestion can play an important role in improving the physiological and psychological parameters of critically ill patients, especially in intensive care units (ICU). Clinical applications of auditory suggestion often include music therapy, white noise, nature sounds, meditation music and audio recordings with subliminal messages. Music therapy is the most common and most researched form of auditory suggestion. In the mid-20th century, music therapy began to be used as an adjunct therapy in the treatment of various psychological and neurological disorders. However, in modern medicine and psychology, the physiological effects of auditory suggestion are being taken more into account. Studies on the use of auditory suggestion, especially in intensive care units, show that this method can increase the hemodynamic stability of patients and reduce their stress levels.

With the sense of hearing, which is the last lost sense of hearing of human beings, the physiological and comfort parameters of the patients can be positively changed by the bed bath given to critically ill patients accompanied by auditory suggestion. Since patients who cannot communicate verbally have no control over themselves and their environment, it is known that talking with these patients has a therapeutic value. Accordingly, the aim of this study was to examine the effect of bed bath given to intensive care unit patients accompanied by auditory suggestion on physiologic and comfort parameters.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Glasgow Coma Scale score: 8 and above
* Richmond Agitation-Sedation Scale (RASS) score between +2 and -3
* APACHE II score <10 points
* Stayed in the ICU for at least 24 hours
* Continues breathing with invasive mechanical ventilation support device
* Not receiving antihypertensive treatment
* Not taking inotropic drugs that directly affect vital signs (esmolol, noradrenaline, dopamine, adrenaline, dopamine, nitrate, etc.)
* No wounds/injuries that would prevent bed bathing
* There is no harm in moving it
* Routine blood gas values (no extra blood gas sample will be taken for this study)

Exclusion Criteria:

* Glasgow Coma Scale score: Under 8
* Richmond Agitation-Sedation Scale (RASS) score of +3 and above, -4 and below
* APACHE II score >10 points
* Stayed in ICU for less than 24 hours
* Referred to another ICU or clinic during the collection of research data
* Intubated in less than 24 hours
* Treatment protocol changed (hypertension and inotrope etc. drugs started)
* Disturbed physiological parameters during bed bathing
* Restricted mobility
* No request for blood gas collection/no blood gas value
* Patients who exit during the study period will be excluded from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Intensive Care Pain Observation Scale | Before bed bath, immediately and 30 minutes after the bed bat
  It is a scale used specifically for the assessment of pain in unconscious patients receiving mechanical ventilation treatment in ICU. The scale consists of four parameters to assess facial expression, body movements, ventilator compliance and muscle tension. Each parameter is scored between 0 and 2. The minimum score is 0 and maximum score is 8. Scores between 0 and 4 show mild to moderate pain and scores between 5 and 8 show severe pain. Since pain is one of the most important markers of comfort, investigators planned to use this scale for criterion-related validity. It is expected that as pain increases, comfort level decreases.
Comfort Behaviors Checklist | Before bed bath, immediately and 30 minutes after the bed bath
  The Comfort Behaviors Checklist consists of 30 behavioral indicators. In addition, Kolcaba suggests that if the list is the only measurement tool that measures comfort, the individual should give a numerical score to pain and comfort so that comfort can be objectively evaluated. Questions 2, 3, 5, 7, 8, 8, 9, 11, 12, 13, 19, 20, 21, 22, 24, 25, 27 are reverse coded. The list is scored on a 4-point Likert scale. When the list is completed, questions that are not applicable to the individual are given 0 points. The total number of questions answered is multiplied by 4 to obtain the possible score. The scores for all questions are calculated by reversing the questions, and the raw comfort score is obtained. Finally, the possible comfort scores are divided by the raw scores to obtain a decimal number. The decimal part of the obtained score is expressed as a two-digit number. The total score is calculated and then standardized to a scale of 0 (lowest comfort) to 120 (highest comfort).
Change in Heart Rate | Baseline (pre-bed bath), immediately post-bed bath, and 30 minutes post-bed bath
  Heart rate (beats per minute) will be measured before bed bath, immediately after, and 30 minutes after.
Change in Systolic and Diastolic Blood Pressure | Baseline, immediately post, and 30 minutes post-intervention
  Systolic and diastolic blood pressure (mmHg) will be measured at three time points: before, immediately after, and 30 minutes after bed bath.
Change in Respiratory Rate | Baseline, immediately post, 30 minutes post
  Respiratory rate (breaths per minute) will be assessed at baseline, immediately after, and 30 minutes after the bed bath.
Change in Body Temperature | Baseline, immediately post, 30 minutes post
  Body temperature (in degrees Celsius) will be recorded at three time points: before, immediately after, and 30 minutes after the bed bath.
Change in Peripheral Oxygen Saturation (SpO₂) | Baseline, immediately post, 30 minutes post
  SpO₂ will be measured using pulse oximetry before and after the bed bath at designated time points.
Change in Blood pH | Baseline, immediately post, 30 minutes post
  Blood pH will be assessed through arterial blood gas sampling at three time points.
Change in Partial Pressure of Oxygen (pO₂) | Baseline, immediately post, 30 minutes post
  pO₂ will be measured through arterial blood gas analysis at three time points.
Change in Partial Pressure of Carbon Dioxide (pCO₂) | Baseline, immediately post, 30 minutes post
  pCO₂ values will be obtained via arterial blood gas analysis at the specified intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No